CLINICAL TRIAL: NCT03098134
Title: The Efficacy of a VR Enhanced Video Exposure Therapy for Dental Phobia - a Randomized Controlled Trial
Brief Title: The Efficacy of a VR Enhanced Video Exposure Therapy for Dental Phobia
Acronym: VR-DENT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ruhr University of Bochum (Other)
Collaborators: Ruhr University of Bochum (Dr. Andre Wannemüller) (Unknown); Zahnklinik Bochum, Augusta Hospital (Prof. Dr. Peter Jöhren) (Unknown); Ruhr University of Bochum (Prof. Dr. Jürgen Margraf) (Unknown)
Responsible Party: Principal Investigator, Dirk Adolph, Head of Clinical Psychophysiology Lab, Ruhr University of Bochum
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VR-DENT-1
Record Dates: First submitted 2017-03-14; First posted 2017-03-31 (Actual); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Dental Phobia
MeSH Terms: interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR-Video-Exposure (Experimental)
  Interventions: Behavioral: Behavior Therapy
- Education-Video- (Active Comparator)
  Interventions: Other: Health Education

INTERVENTIONS:
Behavioral: Behavior Therapy — Virtual Reality and Video based Exposure Therapy
  Arms: VR-Video-Exposure
Other: Health Education — Video based health education covering common myths and false believes about dental surgeries
  Arms: Education-Video-

SUMMARY:
Evaluation of a one session VR - enhanced Video exposure therapy for dental phobia. Diagnosed dental phobics will be randomly assigned to one of two conditions: (1) Psychoeducation + VR exposure (2) Psychoeducation + Video Control treatment. Prior to getting the therapy, participants will be evaluated with a questionnaire battery, diagnosed with a structured clinical interview and will participate in a psychophysiological symptom assessment. Then, after a 2-week waiting period, participants again fill in questionnaires, and the Intervention will take place. Within 2-weeks after the second questionnaire assessment participants will be screened with the structured interview again and will fill in questionnaires.

ELIGIBILITY:
Inclusion Criteria:

- diagnosed Specific Dental Phobia

Exclusion Criteria:

* Schizophrenia or other Psychotic Illnesses
* Bipolar Disorder
* Chronic Headache
* other neurological disorders such as epilepsy
* Hearing problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-04 (Estimated); Primary Completion 2017-12-31 (Estimated); Study Completion 2018-05-01 (Estimated)

PRIMARY OUTCOMES:
Change in Subjective Dental Anxiety | 4 month
  Assessed at time 0 (at inclusion) 1 (pre therapy, two weeks after inclusion), 2(post therapy, 2 weeks after time 1) and at follow up (4 month after time 0) with Dental Anxiety Scale (DAS, 4-item scale, range 4-20)
Change in Dysfunctional Dental Cognitions | 4 months
  Assessed with Dental Cognition Questionnaire (DCQ, 38 dichotomous items, range 0-38) Assessed at time 0 (at inclusion), time 1 (pre therapy, two weeks after time 0), time 2 (post therapy, 2 weeks after time 1) and at follow up (4 month after time 0)

SECONDARY OUTCOMES:
Change in Psychophysiological defensive reactivity | 4 weeks
  Participants will take part in a passive Picture viewing paradigm. They will be exposed to dental anxiety related Pictures, generally negative pictures, neutral, and positive pictures. Outcome measures will be withdrawal-related motor responding (assessed with the startle-reflex), as well as heart frequency change towards the pictures, The task will be applied at inclusion (time 0) and post therapy (4 weeks after inclusion)

OTHER OUTCOMES:
Change in dental avoidance behavior | within three month after the therapy took place
  Each participant will be asked to arrange an appointment in a cooperating dental Hospital. It will be assessed (1) if participant makes a - (2) and attends to - first appointment (3) if participant tolerates oral inspection and dental treatment (4) how many further appointments will be made

IPD SHARING:
Plan to Share IPD: No